CLINICAL TRIAL: NCT06090760
Title: Mindfulness Intervention on Wellbeing During OSN
Brief Title: Mindfulness Intervention and Online Social Networking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GU Mingyue Michelle, Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EduUHK01
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-05

CONDITIONS: Mindfulness
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: waitlist control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Intervention Group (Experimental): Mindfulness training will be provided to the participant after randomization for dealing with social media use.
  Interventions: Behavioral: Mindfulness
- Waitlist Control Group (No Intervention): No mindfulness training will be provided to the participants.

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness is "paying attention in a particular way: on purpose, in the present moment, and non-judgmentally" (Kabat-Zinn 1994, 4) and has five facets: awareness, nonjudgement, nonreactive, observe, and describe (Baer et al., 2006).
  Arms: Mindfulness Intervention Group

SUMMARY:
This study aims to examine (a) the effects of mindfulness-based intervention on wellbeing including psychological, social, and emotional wellbeing, depressive symptoms, and stress and (b) the extent to which demographics, OSN use, and mindfulness mediate these effects.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old

Exclusion Criteria:

* have not complete the application form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Social Media Engagement | 8 weeks
  The Social Media Engagement Scale
Well-being | 8 weeks
  Well-being Scale
Emotion | 8 weeks
  Difficulties in Emotion Regulation Scale
Depression | 8 weeks
  Depression and Anxiety Stress Scales

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gu, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- Ngar-sze Lau, Hong Kong, Hong Kong